CLINICAL TRIAL: NCT00101517
Title: Partnership Programs to Reduce Cardiovascular Disparities - Morehouse-Emory Partnership
Brief Title: Partnership Programs to Reduce Ethnic Differences in the Risk of Cardiovascular Disease
Acronym: META-HEALTH
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Principal Investigator, Emory University
Other Study IDs: IRB00024856a; U01HL079156 (NIH); U01HL079214 (NIH); 1284 (Other: Other)
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity; Metabolic Syndrome X
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to improve cardiovascular disease (CVD) outcomes in racial and ethnic minorities. Specifically, the study seeks to systematically characterize potential ethnic differences in obesity-related CVD by drawing upon the fields of psychology, physiology, biochemistry, nursing, and clinical medicine.

DETAILED DESCRIPTION:
BACKGROUND:

While there has been great progress in reducing CVD morbidity and mortality in the U.S. over the past 40 years, some minority groups have not shared fully in this progress and continue to have lower life expectancy and higher CVD morbidity. On average, minorities have less access to medical care, receive less aggressive care and fewer diagnostic and therapeutic cardiac procedures, and adhere poorly to prescribed medical regimens. Thus, research to reduce health disparities by improving CVD outcomes in minorities offers potential for a substantial positive public heath impact. Academic medical centers and institutions capable of carrying out such research, however, often lack access to and the trust of minority patients. Minority patients often receive fragmented care because they lack access to regular medical care, present to emergency departments rather than primary care physicians for complications of an advanced chronic CVD condition, and are less likely to follow medical regimens. Minority communities often harbor distrust of clinical research. Minority patients report greater satisfaction when receiving care from minority providers and are reluctant to receive treatment outside their minority healthcare serving systems.

In general, minorities have high rates of hypertension, elevated cholesterol, cigarette smoking, obesity, metabolic syndrome, and diabetes, as well as other behavioral, environmental, and occupational risk factors for cardiovascular diseases, such as sleep problems - all elements that contribute to excess CVD morbidity and mortality. The causes of minority health disparities are complex and incompletely understood. Although evidence of genetic, biologic, and environmental factors is well documented, poor outcomes are also attributed to under-treatment. Such under-treatment may be due to limited access to health care or, in some cases, break-down of the medical system, or failure of the physician and/or patient to allow for optimal health care, even when access is not impaired. The complex interactions of behavior, socio-economic status (SES), culture, and ethnicity are important predictors of health outcomes and sources of health disparities. Despite efforts to elucidate genetic and environmental risk factors and to promote cardiovascular health in high-risk populations, trends in CVD outcomes suggest that CVD health disparities continue to widen.

The Partnerships Program to Reduce Cardiovascular Health Disparities involves collaboration between research-intensive medical centers (RIMCs) that have a track record of NIH-supported research and patient care and minority healthcare serving systems (MSSs) that lack a strong research program. Each Partnership Program will: a) design and carry out multiple interdisciplinary research projects that investigate complex biological, behavioral,and societal factors that contribute to CVD health disparities and facilitate clinical research within the MSS to improve CVD outcomes and reduce health disparities, and b) provide reciprocal educational and skills development programs so that investigators will be able to conduct research aimed at reducing cardiovascular disparities and thereby enhance research opportunities, enrich cultural sensitivity, and improve cardiovascular research capabilities at both institutions.

The Request for Applications for Partnership Programs to Reduce Cardiovascular Disparities was released in September 2003. The awards were made in September 2004.

DESIGN NARRATIVE:

Over the past decade, there has been an explosive increase in obesity among all age groups within the U.S. population. This epidemic is particularly problematic among African Americans in the Southeast. Although genetic factors play a contributory role, it is postulated that ethnic disparities in obesity and obesity-related CVD are related to a dynamic interplay between biological factors and the behavioral response to the unique environmental context within ethnic communities. Obesity is often associated with perturbations in the metabolic and physiologic milieu. A cluster of obesity-related abnormalities has been defined as the "Metabolic Syndrome". The CVD complications of obesity appears to be related to the capacity for adipose tissue itself to generate "adipokines" that directly predispose to insulin-resistance, endothelial dysfunction, inflammation, and vascular disease.

The study will use state-of-the-art approaches to define potential ethnic differences in the profile of metabolic, physiologic, and biochemical features associated with obesity as well as the salutary responses to lifestyle modification. The program uses a multi-disciplinary strategy to systematically characterize potential ethnic differences in obesity-related CVD by drawing upon the fields of psychology, physiology, biochemistry, nursing, and clinical medicine. In a thematic series of inter-related studies, the program's research plan ranges from epidemiology studies within the ethnic communities, to patient-centered clinical trial interventions within ethnic community practices, to the analysis of novel biomarkers of human pathobiology. This collaborative multi-investigator team is built upon a complementary partnership between the Morehouse School of Medicine and Emory University. This partnership shares a joint commitment to address the striking ethnic disparities in the high-risk CVD population. The specific aims are: 1) to define the relative influence of psychosocial/cultural factors and biological mediators as determinants of ethnic disparities in obesity and the metabolic syndrome in a population-based bi-racial cohort; 2) to define the effectiveness of patient-targeted behavioral interventions to enhance the health of African American patients with the Metabolic Syndrome in the context of community-based clinical practices; 3) to assess the impact of innovative lifestyle intervention strategies on conventional and novel biomarkers of vascular disease risk in African Americans; and 4) to enhance the education/training of fellows/practitioners engaged in CVD disparities research/practice and promote partnerships that enhance cardiovascular health within ethnic communities.

ELIGIBILITY:
* African-American or White residents of the metro Atlanta area
* aged 30-78 years

Ages: 30 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African-American and white residents in the metro Atlanta area (Cobb, DeKalb, Fulton, Gwinnett counties) aged 30-78 years
Sampling Method: Probability Sample
Enrollment: 4024 (Actual)
Dates: Start 2004-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Gibbons, Principal Investigator — Morehouse School of Medicine; Arshed Quyyumi, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University School, Atlanta, Georgia